CLINICAL TRIAL: NCT03686865
Title: Peri-implant Marginal Bone and Soft Tissue Conditions Around Single Laser-Lok Implants Placed in Regenerated Extraction Sockets and in Native Bone: A 2-years Results of RCT
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Renzo Guarnieri, adjunct professor, University of Roma La Sapienza
Other Study IDs: 4597 bis
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Partially Edentulous Maxilla, Partially Edentulous Mandible
Keywords: regenerated bone, native bone, dental implant
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dental implants
  Interventions: Device: dental implants

INTERVENTIONS:
Device: dental implants — extraction sockets regenerated with xenograft
  Other Names: porcine derived bone

SUMMARY:
The aim of present study was to compare peri-implant marginal bone loss and soft tissues conditions around single Laser-Lok implants placed in alveolar

DETAILED DESCRIPTION:
Records of 20 consecutive patients treated with dental implants placed in post-extraction sockets augmented with porcine derived bone and 20 consecutive patients with implants placed in native bone were reviewed. For each implant, the radio- graphs from the surgical appointment were compared to those from the last follow-up visit and evaluated regarding changes of marginal bone level over time.

ELIGIBILITY:
Inclusion Criteria:

* mono-edentulism, age ≥ 18 years, good general health, without contraindications to implant surgery

Exclusion Criteria:

* lack of a periodontal chart and periapical radiograph at the beginning and at the end of follow-up period, alcohol and drug abuse, pregnancy, or uncontrolled metabolic disorders, tobacco smoking (> 10 cigarettes/day), full mouth plaque score (FMPS), and full mouth bleeding score /FMBS) ≥25%, teeth adjacent to the implant area (mesial and distal) affected by untreated periodontal and/or endodontic infections.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with monoedentulism
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
peri-implant marginal bone loss | 2 years

SECONDARY OUTCOMES:
peri-implant soft tissue conditions | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Universita la Sapienza, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Carlsson GE, Bergman B, Hedega ̊rd B. Changes in contour of the maxillary alveolar process under im- mediate dentures. A longitudinal clinical and x-ray cephalometric study covering 5 years. Acta Odontol Scand 1967;25:45-75. 2. Arau ́jo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol 2005;32:212-218. 3. Pietrokovski J, Massler M. Alveolar ridge resorption following tooth extraction. J Prosthet Dent 1967;17: 21-27. 4. Johnson K. A study of the dimensional changes occurring in the maxilla following tooth extraction. Aust Dent J 1969;14:241-244. 5. Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: A clinical and radiographic 12- month prospective study. Int J Periodontics Restor- ative Dent 2003;23:313-323. 6. Arau ́jo MG, Carmagnola D, Berglundh T, Thilander B, Lindhe J. Orthodontic movement in bone defects augmented with Bio-Oss. An experimental study in dogs. J Clin Periodontol 2001;28:73-80. 7. Carmagnola D, Berglundh T, Lindhe J. The effect of a fibrin glue on the integration of Bio-Oss with bone tissue. An experimental study in Labrador dogs. J Clin Periodontol 2002;29:377-383. 8. Cardaropoli G, Arau ́jo M, Hayacibara R, Sukekava F, Lindhe J. Healing of extraction sockets and surgically produced - augmented and non-augmented - defects in the alveolar ridge. An experimental study in the dog. J Clin Periodontol 2005;32:435-440. 9. Becker W, Clokie C, Sennerby L, Urist MR, Becker BE. Histologic findings after implantation and evaluation of different grafting materials and titanium micro screws into extraction sockets: Case reports. J Periodontol 1998;69:414-421. 10. Artzi Z, Tal H, Dayan D. Porous bovine bone mineral in healing of human extraction sockets. Part 1: Histo- morphometric evaluations at 9 months. J Periodontol 2000;71:1015-1023. 11. Artzi Z, Tal H, Dayan D. Porous bovine bone mineral in healing of human extraction sockets: 2. Histochemical observations at 9 months. J Periodontol 2001;72:152- 159. 12. Iasella JM, Greenwell H, Miller RL, et al. Ridge preservation with freeze-dried bone allograft and a col- lagen membrane compared to extraction alone for implant site development: A clinical and histologic study in humans. J Periodontol 2003;74:990-999. 13. Carmagnola D, Adriaens P, Berglundh T. Healing of human extraction sockets filled with Bio-Oss. Clin Oral Implants Res 2003;14:137-143. 14. Becker W, Urist M, Becker BE, et al. Clinical and histologic observations of sites implanted with intrao- ral autologous bone grafts or allografts. 15 human case reports. J Periodontol 1996;67:1025-1033. 15. Froum S, Cho SC, Rosenberg E, Rohrer M, Tarnow D. Histological comparison of healing extraction sockets implanted with bioactive glass or demineralized freeze-dried bone allograft: A pilot study. J Periodontol 2002;73:94-102. 16. Barone A, Aldini NN, Fini M, Giardino R, Calvo Guirado JL, Covani U. Xenograft versus extraction alone for ridge preservation after tooth removal: A clinical and histomorphometric study. J Periodontol 2008;79:1370-1377. 17. Lekovic V, Kenney EB, Weinlaender M, et al. A bone regenerative approach to alveolar ridge maintenance following tooth extraction. Report of 10 cases. J Periodontol 1997;68:563-570. 18. Lekovic V, Camargo PM, Klokkevold PR, et al. Pres- ervation of alveolar bone in extraction sockets using bioabsorbable membranes. J Periodontol 1998;69: 1044-1049. 19. Nevins M, Camelo M, De Paoli S, et al. A study of the fate of the buccal wall of extraction sockets of teeth with prominent roots. Int J Periodontics Restorative Dent 2006;26:19-29. 20. Albrektsson T, Bra ̊ nemark PI, Hansson HA, Lindstro ̈ m J. Osseointegrated titanium implants. Requirements for ensuring a long-lasting, direct bone-to-implant anchorage in man. Acta Orthop Scand 198